CLINICAL TRIAL: NCT00474604
Title: MRI Evaluation of Breast Tumor Growth and Treatment Response
Brief Title: Breast MRI in Women With Known or Suspected Breast Cancer and in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Professor; Radiation Oncology, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC BRE 0588; P30CA068485 (NIH); VU-VICC-BRE-0588; VU-VICC-IRB-051230
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants without breast cancer (Active Comparator)
  Interventions: Procedure: diffusion-weighted magnetic resonance imaging; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: magnetic resonance spectroscopic imaging
- Participants with breast cancer (Experimental)
  Interventions: Procedure: diffusion-weighted magnetic resonance imaging; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: magnetic resonance spectroscopic imaging

INTERVENTIONS:
Procedure: diffusion-weighted magnetic resonance imaging — A scan will be performed.
Procedure: dynamic contrast-enhanced magnetic resonance imaging — A scan will be performed.
Procedure: magnetic resonance spectroscopic imaging — A scan will be performed.

SUMMARY:
RATIONALE: Diagnostic procedures, such as MRI, may help diagnose breast cancer. It may also help doctors predict a patient's response to treatment.

PURPOSE: This clinical trial is studying breast MRI in women with known or suspected breast cancer and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and combine advanced, quantitative, multiparametric magnetic resonance imaging methods (i.e., dynamic contrast-enhanced MRI [DCE-MRI], diffusion-weighted MRI [DW-MRI], and magnetic resonance spectroscopy [MRS]) to characterize breast tumors in women with known or suspected breast cancer.
* Identify surrogate biomarkers that can guide diagnosis and treatment of breast cancer using these methods.
* Correlate biochemical information obtained from magnetic resonance analysis with clinical, radiologic, and pathologic findings in these patients.
* Establish an imaging data bank that includes information on DCE-MRI, DW-MRI, and MRS findings in these patients and in healthy participants.

OUTLINE: Quantitative, multi-parametric magnetic imaging methods will be employed for breast imaging for the following subjects:

* Group A: Healthy volunteers who undergo up to 3 breast MRIs over 6 weeks.
* Group B: Patients diagnosed with breast cancer who will: 1) undergo preoperative breast MRI followed by definitive surgery or 2) undergo MRI prior to initiating neoadjuvant chemotherapy, at 1-2 weeks after initiation of chemotherapy, and prior to definitive surgery.

Clinical information, including radiologic and pathologic data, on all patients is collected for inclusion in the imaging data bank.

After completion of the study, patients and healthy participants are followed periodically.

ELIGIBILITY:
Inclusion criteria:

Women who satisfy the following conditions are the only subjects who will be eligible for this study:

* Normal volunteers
* Subjects with known or suspected breast disease
* Subjects must have signed an approved consent form.
* Subjects must be ≥ 18 years old.
* The protocol nurse will check with the patient that there is no h/o kidney disease
* Normal creatinine and estimated GFR* within 30 days under the following circumstances

  * Had abnormal creatinine in the last 60 days
  * Are over 60 years of age
  * Has received chemotherapy within the past 30 days
  * Has diabetes, HIV, renal disease or hx of renal cancer
* * GFR will be calculated using: http://www.kidney.org/professionals/kdoqi/gfr_calculator.cfm
* Patients with an eGFR>90ml/min reported within 30 days, and who have not had intervening chemotherapy or other treatment or condition that might deteriorate renal function, may receive any gadolinium agent.

Exclusion Criteria:

* Children will be excluded from this study.
* Pregnant women and women who are breast feeding will be excluded from this study. (The Vanderbilt University Medical Center radiology "MRI Procedure Screening Form" will be used to identify and exclude subjects who are pregnant or breastfeeding. A urine pregnancy test/or serum beta HCG will also be performed for each pre-menopausal subject.)
* Subjects found to have any constitutionally present non-MR compatible ferromagnetic materials will be excluded from this study.
* Patients who are acutely ill who are deemed by their treating physician as not suitable candidates for this study
* Subjects for whom an MRI is technically not feasible (e.g. breast volume, obesity)
* Subjects who have vascular access ports or other implanted devices rated as anything other than "Safe" or "Conditional 6"

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of advanced, quantitative, multi-parametric magnetic resonance imaging (MRI) methods for characterizing breast tumors to develop potential surrogate imaging markers for diagnosis and prediction of treatment response | on-study date and at 6 months, up to 4 years
  Quantitative, multi-parametric MRI imaging methods include Dynamic Contrast MRI, Diffusion Weighted MRI, and Magnetic Resonance Spectroscopy. Patients will include healthy female volunteers and women diagnosed with breast cancer. Time frames begin at study entry (healthy volunteers) , pre-surgical and pre- and post-chemotherapy (breast cancer patients)

SECONDARY OUTCOMES:
Correlation of biochemical data obtained from magnetic resonance analysis with clinical, radiological, and pathological findings | at 6 months
  Biochemical data from advanced MRIs are compared and contrasted with findings from patients' clinical, chemotherapeutic, and radiologic treatments for breast cancer.
Establishment of an imaging data bank | at 6 months
  Results of advanced MRI imaging methods for subjects assessed after completion of all MRI procedures

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Yankeelov TE, Lepage M, Chakravarthy A, Broome EE, Niermann KJ, Kelley MC, Meszoely I, Mayer IA, Herman CR, McManus K, Price RR, Gore JC. Integration of quantitative DCE-MRI and ADC mapping to monitor treatment response in human breast cancer: initial results. Magn Reson Imaging. 2007 Jan;25(1):1-13. doi: 10.1016/j.mri.2006.09.006. Epub 2006 Nov 21. PMID 17222711
- [Derived] Li X, Abramson RG, Arlinghaus LR, Chakravarthy AB, Abramson V, Mayer I, Farley J, Delbeke D, Yankeelov TE. An algorithm for longitudinal registration of PET/CT images acquired during neoadjuvant chemotherapy in breast cancer: preliminary results. EJNMMI Res. 2012 Nov 16;2(1):62. doi: 10.1186/2191-219X-2-62. PMID 23157877
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/